CLINICAL TRIAL: NCT07097051
Title: Multi-session Transcranial Alternating Current Stimulation to Improve Dual-task Standing and Brain Activity in Older Adults With Mild Cognitive Impairment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: High Point University (Other)
Collaborators: Wake Forest University Health Sciences (Other); Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Melike Kahya, Assistant Professor, High Point University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-FY2025-70
Record Dates: First submitted 2025-07-21; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: brain stimulation; balance; cognition; executive function
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tACS (Experimental): The investigators will administer the transcranial alternating current stimulation (tACS) intervention individually tailored to peak alpha power to the participants. This intervention will utilize 8 electrodes; electrode placement and current parameters for each electrode have been optimized using a standard brain to generate an average electric field of 0.25 V/m. To ensure adherence to current safety recommendations for tACS, optimizations will be constrained to a maximum of total injected current 4.0 mA and a max. current per electrode of 2.0 mA. Stimulation will start and end with a 60 s ramp up/down to maximize comfort and the entire session will take 22-minute. This standard approach is both well-tolerated and safe in older adults.
  Interventions: Other: real tACS
- sham tACS (Placebo Comparator): The investigators will administer the sham tACS intervention to the participants. They will use an active sham in which very low-level alternating currents (0.5 mA total) will be transferred between electrodes in close proximity on the scalp throughout the session. Stimulation will start and end with a 60 s ramp up/down to maximize comfort and the entire session will last in 22-minutes.
  Interventions: Other: sham tACS

INTERVENTIONS:
Other: real tACS — Those who randomized into real tACS arm will receive ten-session of individually tailored tACS targeting peak alpha power for 20-minutes
  Arms: real tACS
Other: sham tACS — Those who randomized into sham tACS arm will receive ten-session of active sham tACS intervention for 20-minutes
  Arms: sham tACS

SUMMARY:
Older adults with Mild Cognitive Impairment (MCI) often show less brain activity in a specific range (8-13 Hz, known as alpha power) compared to healthy older adults. Those with lower alpha activity, especially in the front part of the brain, usually have problems with executive functions like planning and multitasking. Our research has shown that older adults with lower alpha power in these areas also struggle more with balance when they have to do two things at once (like standing and performing a cognitive task simultaneously).

The investigators believe that increasing alpha power in older adults with MCI could improve their balance and executive function, helping them stay independent longer. In early studies, the investigators found that using transcranial alternating current stimulation (tACS) at 10 Hz on the front part of the brain can boost alpha power and balance immediately after a single session in older adults with MCI. The effect was stronger in those whose natural brain activity was close to the 10 Hz stimulation.

Based on these findings, the investigators plan to conduct a pilot study with older adults aged 65-85 years with MCI. Participants will be randomly assigned to receive either real tACS or a sham (placebo) treatment. Our main hypothesis is that real tACS will improve balance when multitasking, and these improvements will last for 1 to 3 months after the treatment. The investigators also believe that tACS will enhance other aspects of executive function and mobility and that these improvements will be linked to increased alpha activity in the brain.

Through this study, we aim to gather strong evidence that tailored tACS is a promising treatment to improve cognitive and motor functions and overall brain activity in older adults with MCI.

DETAILED DESCRIPTION:
Older adults with Mild Cognitive Impairment (MCI) exhibit reduced brain alpha power (i.e., activity fluctuations in the 8-13 Hz range) compared to healthy older adults, and older adults who exhibit lower alpha activity in the fronto-central areas tend to have impaired executive function. In addition, our group has demonstrated that older adults who exhibit lower fronto-central alpha power during dual-task standing (i.e., standing while performing an unrelated cognitive task) have worse standing balance performance. We, therefore, contend that strategies designed to increase alpha power in older adults with MCI hold promise to enhance dual-task balance and other measures of executive function, and ultimately help these vulnerable individuals maintain functional independence over time.

In our preliminary studies, we have demonstrated that a single exposure to transcranial alternating current stimulation (tACS) delivered at 10 Hz over the fronto-central regions of the brain increases alpha power and dual-task balance in older adults with MCI, when tested just after stimulation. We have also observed that in older adults with MCI, 10 Hz tACS appears to have a greater effect on alpha activity and dual-task balance in those individuals whose peak alpha frequency happens to be at or near the stimulation frequency (10 Hz).

Given the above evidence, we will conduct a pilot, double-blinded, parallel-arm, randomized controlled trial in ambulatory women and men aged 65-85 years with MCI. Our primary hypothesis is that compared to sham, tACS will improve dual-task balance when tested at the end of the intervention, and that such effects will persist at the 1- and 3-month follow-up. We further hypothesize that 1) tACS, compared to sham, will improve performance in other clinically-tractable measures of executive function and mobility, and 2) that tACS-induced improvements in dual-task balance will correlate with increased alpha brain activity. Through these efforts, we anticipate providing rigorous preliminary data that individually-tailored tACS is an effective therapeutic option capable of inducing sustained improvements in cognitive-motor functions, as well as underlying brain activity, in older adults with MCI.

ELIGIBILITY:
Inclusion Criteria:

* Age 65+
* Who have been diagnosed with cognitive impairment (based in MoCA or TICS and Clinical Dementia Rating: CDR 0.5)
* Ability to stand and walk independently
* Willing and capable to give informed consent for the participation in the study after it has been thoroughly explained
* Cut off of MOCA score >18 will be applied
* Able and willing to comply with all study requirements informed consent form was signed
* Understanding of the ICF will be assessed by asking the participant to answer the following three questions: 1) What is the purpose of this study? 2) What are the risks of study involvement? 3) If you decide to participate, are you allowed to withdraw from the study at any time? Answers will be recorded by study personnel on the "Assessment of Protocol Understanding" form (see attached). Insufficient understanding will be defined by one or more incorrect answers, as determined at the discretion of the investigator.

Exclusion Criteria:

* Cut off of MOCA score <18 will be applied
* Major psychiatric co-morbidity including major depressive disorder, schizophrenia or psychosis
* Blindness or other disabilities that prevent task performance
* Self-reported history of stroke or neurodegenerative disorders other than MCI.
* Self-reported active cancer for which chemo-/radiation therapy is being received.
* Contraindications to tACS, as recorded on a standardized screening questionnaire, which include a reported seizure within the past two years, use of neuro-active drugs, self-reported presence of specific implanted medical devices (e.g., deep brain stimulator, medication infusion pump, cochlear implant, pacemaker, etc.), or the presence of any active dermatological condition, such as eczema, on the scalp.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
EEG alpha-band power | Baseline, immediate post-intervention assessments, Follow-up visit #1 (4 weeks later of post-intervention assessment, Follow-up visit #2 (12 weeks later post-intervention assessment).
  Change of EEG oscillations and frequency coupling at 8-13 Hz
Change of postural sway speed | Baseline, immediate post-intervention assessments, Follow-up visit #1 (4 weeks later of post-intervention assessment, Follow-up visit #2 (12 weeks later post-intervention assessment).
  his metric assesses the ability to control standing posture

SECONDARY OUTCOMES:
Change of executive function score | Baseline, immediate post-intervention assessments, Follow-up visit #1 (4 weeks later of post-intervention assessment, Follow-up visit #2 (12 weeks later post-intervention assessment).
  This metric reflects measures of executive function scores based on individual neuropsychological test of Trail-making Test B completion time
Change of dual-task gait speed | Baseline, immediate post-intervention assessments, Follow-up visit #1 (4 weeks later of post-intervention assessment, Follow-up visit #2 (12 weeks later post-intervention assessment).
  This metric (m/s) assesses the ability to walk and perform a cognitive task at the same time and predicts cognitive decline and the development of dementia.
Timed Up and Go Test completion time | Baseline, immediate post-intervention assessments, Follow-up visit #1 (4 weeks later of post-intervention assessment, Follow-up visit #2 (12 weeks later post-intervention assessment).
  This test assesses time to complete standing from a chair, walking three meters, turning around a cone and returning to a seated position in the chair.
Short Physical Performance Battery score | Baseline, immediate post-intervention assessments, Follow-up visit #1 (4 weeks later of post-intervention assessment, Follow-up visit #2 (12 weeks later post-intervention assessment).
  This common test assesses physical functioning. The score is ranging from 0 to 12, with higher scores indicating better physical performance.
Montreal Cognitive Assessment (MoCA) | Baseline, immediate post-intervention assessments, Follow-up visit #1 (4 weeks later of post-intervention assessment, Follow-up visit #2 (12 weeks later post-intervention assessment).
  This common test assesses global cognitive function. The Montreal Cognitive Assessment (MoCA) test is scored out of a total of 30 points, with higher scores indicating better cognitive function.
Dual-task Standing Postural Sway Path | Baseline, immediate post-intervention assessments, Follow-up visit #1 (4 weeks later of post-intervention assessment, Follow-up visit #2 (12 weeks later post-intervention assessment).
  This metric assesses the ability to stand and perform a cognitive task at the same time and predicts cognitive decline and the development of dementia.
Serial subtraction test performance | Baseline, immediate post-intervention assessments, Follow-up visit #1 (4 weeks later of post-intervention assessment, Follow-up visit #2 (12 weeks later post-intervention assessment).
  This metric assesses the number of correct response on serial subtraction test while standing
Digit Span total recall | Baseline, immediate post-intervention assessments, Follow-up visit #1 (4 weeks later of post-intervention assessment, Follow-up visit #2 (12 weeks later post-intervention assessment).
  This metric assesses working memory.
WAIS-IV Coding test completion time | Baseline, immediate post-intervention assessments, Follow-up visit #1 (4 weeks later of post-intervention assessment, Follow-up visit #2 (12 weeks later post-intervention assessment).
  This metric assesses sustained attention and motor speed.
Brain networks connectivity changes | Baseline and immediate post-intervention assessments
  Measures of functional brain connectivity based on resting-state functional magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- High Point University, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No